CLINICAL TRIAL: NCT01706250
Title: U0289-401: An Evaluator Blinded, 8 Week, Split-Face Study to Evaluate and Compare the Efficacy and Tolerability of MAXCLARITY II and PROACTIV in Subjects With Acne
Brief Title: U0289-401: Eight Week, Split-face, Study to Determine and Compare the Efficacy and Tolerability of MAXCLARITY™ II to PROACTIV™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 114550
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Salicylic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MAXCLARITY II (Experimental): MaxClarity II (2.5% BPO) Foam Cleanser and Foam Treatment and (0.5% Salicylic Acid) Toner Foam. Available over the counter. Each subject applies both arms (MaxClarity II and Proactiv) simultaneously for the entire duration of the study (8 weeks), each arm to be applied to one side of the face only (split-face study) according to randomization.
  Interventions: Other: MAXCLARITY II (2.5% BPO) Foam Cleanser; Other: MAXCLARITY II (2.5% BPO) Foam Treatment; Other: MAXCLARITY II (0.5% Salicylic Acid) Toner Foam
- PROACTIV (Active Comparator): Proactiv (2.5% BPO) Renewing Cleanser and Repairing Lotion and Revitalizing Toner. Available over the counter. Each subject applies both arms (MaxClarity II and Proactiv) simultaneously for the entire duration of the study (8 weeks), each arm to be applied to one side of the face only (split-face study) according to randomization.
  Interventions: Other: PROACTIV (2.5% BPO) Renewing Cleanser; Other: PROACTIV (2.5% BPO) Repairing Lotion; Other: PROACTIV (2.5% BPO) Revitalizing Toner

INTERVENTIONS:
Other: MAXCLARITY II (2.5% BPO) Foam Cleanser — Available over the counter.
  Arms: MAXCLARITY II
Other: MAXCLARITY II (2.5% BPO) Foam Treatment — Available over the counter.
  Arms: MAXCLARITY II
Other: MAXCLARITY II (0.5% Salicylic Acid) Toner Foam — Available over the counter.
  Arms: MAXCLARITY II
Other: PROACTIV (2.5% BPO) Renewing Cleanser — Available over the counter.
  Arms: PROACTIV
Other: PROACTIV (2.5% BPO) Repairing Lotion — Available over the counter.
  Arms: PROACTIV
Other: PROACTIV (2.5% BPO) Revitalizing Toner — Available over the counter.
  Arms: PROACTIV

SUMMARY:
One of the main success factors in acne therapy is user compliance with treatment, product cost, availability and ease of use. Poor compliance may translate into decreased efficacy (either not improving symptoms well enough or not improving symptoms fast enough), tolerability issues or adverse effects (eg, erythema, dryness, or peeling of the skin), a lack of understanding of the instructions for use, or product cost/availability. Whatever the reason, poor compliance translates to decreased efficacy and increased frustration on the part of the user.

The current study will evaluate and compare the efficacy and tolerability of 2 over-the-counter, topical benzoyl peroxide (BPO) product lines in subjects with acne: MAXCLARITY II (2.5% BPO) Foam Cleanser and Foam Treatment and (0.5% Salicylic Acid) Toner Foam compared with PROACTIV (2.5% BPO) Renewing Cleanser and Repairing Lotion and Revitalizing Toner.

DETAILED DESCRIPTION:
Acne vulgaris is an extremely common dermatological disease that is found typically in adolescence and young adulthood. Acne vulgaris manifests with open and closed comedones (blackheads and whiteheads), papules, pustules, nodules, and cysts on the face, neck, and trunk. Scarring can occur, particularly if the lesions are inflamed and deep, even in the absence of external manipulation (eg, picking and squeezing) of the skin.

Acne vulgaris can be treated with a variety of agents that are selected to address the pathogenic factors assumed to be responsible for the type and degree of manifested acne lesions. Monotherapy and combination therapy regimens are both useful. Topical agents are generally used as first-line therapy and include retinoids, antibiotic preparations (eg, erythromycin and clindamycin), benzoyl peroxide (BPO), alpha and beta hydroxy acids (eg, glycolic and salicylic acid preparations), and azelaic acid. Systemic therapies are initiated in patients with moderate to severe inflammatory acne that does not respond to topical therapy.

Benzoyl peroxide has antimicrobial and anti inflammatory properties and is often considered an important component of acne treatment. Benzoyl peroxide is frequently the first product that adolescents will use for acne because it can be purchased without a prescription in several different concentrations and formulations.

One of the main success factors in acne therapy is user compliance with treatment, product cost, availability and ease of use. Poor compliance may translate into decreased efficacy (either not improving symptoms well enough or not improving symptoms fast enough), tolerability issues or adverse effects (eg, erythema, dryness, or peeling of the skin), a lack of understanding of the instructions for use, or product cost/availability. Whatever the reason, poor compliance translates to decreased efficacy and increased frustration on the part of the user.

The current study will evaluate and compare the efficacy and tolerability of 2 common, over-the-counter, topical benzoyl peroxide (BPO) product lines in subjects with acne: MAXCLARITY II (2.5% BPO) Foam Cleanser and Foam Treatment and (0.5% Salicylic Acid) Toner Foam compared with PROACTIV(2.5% BPO) Renewing Cleanser and Repairing Lotion and Revitalizing Toner.

This is a randomized, 2 center, evaluator-blinded, split-face efficacy and tolerability study of MAXCLARITYII and PROACTIV, 2 over-the-counter, topical benzoyl peroxide product lines, in subjects with acne. Approximately 40 subjects, aged from 16 to 29 years, inclusive, with mild facial acne vulgaris are expected to participate in the study. No more than 50% of the subjects at each site can be enrolled under the age of 20.

An expert grader (blinded evaluator) will complete counts of inflamed lesions (papules/pustules) and noninflamed lesions (open/closed comedones), the Investigator's Static Global Assessment (ISGA), and an assessment of tolerability of each side of the face at each study visit. Subjects will assess tolerability on each side of the face at each study visit and will complete a product acceptability and preference questionnaire at the end of the study.

The study duration will be 8 weeks (56 days) with visits at baseline (day 1), week 1m week 2, week 4 and week 8. Only the expert grader (evaluator) will be blinded to the study product assignments; subjects and study nurses/coordinator will not be blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed.
2. Male or female aged from 16 to 29 years, inclusive, at time of consent. No more than 50% of the subjects at each site can be enrolled under the age of 20.
3. Mild facial acne vulgaris, characterized by at least 12 facial inflammatory lesions (papules and pustules) and/or noninflammatory lesions (open and closed comedones) on the face.
4. Able to complete the study and to comply with study instructions.
5. Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses. Acceptable contraceptive methods include the following:

   * Hormonal contraception, including oral, injectable, or implantable methods started at least 2 months prior to screening. If hormonal contraception was started less than 2 months prior to screening, then a form of nonhormonal contraception should be added until the third continuous month of hormonal contraception has been completed.
   * Two forms of reliable nonhormonal contraception, to include the use of either an intrauterine device plus a reliable barrier method or 2 reliable barrier methods. Reliable barrier methods include condoms or diaphragms. A cervical cap is also a reliable barrier method, provided that the female subject has never given birth naturally. The combined use of a condom and spermicide constitute 2 forms of acceptable nonhormonal contraception, provided that they are both used properly. The use of spermicide alone and the improper use of condoms are inferior methods of contraception. Subjects with surgical sterilization, including tubal sterilization or partner's vasectomy, must use a form of nonhormonal contraception. A barrier method or sterilization plus spermatocide is acceptable.
   * Women who are not currently sexually active must agree to use a medically accepted method of contraception should she become sexually active while participating in the study.

Exclusion Criteria:

1. Female who is pregnant, trying to become pregnant, or breast feeding.
2. Has active or chronic skin allergies.
3. Has a history of acute or chronic disease that might interfere with or increase the risk of study participation.
4. Had skin cancer treatment in preceding 12 months.
5. Has damaged skin on facial areas (eg, sunburn, tattoo, or scar)
6. Had any medical procedure (eg, laser resurfacing, chemical peel, or plastic surgery) on facial areas in preceding 12 months.
7. Had any cosmetic procedure (eg, microdermabrasion) on facial areas within 8 weeks of the baseline visit.
8. Has any dermatological disorder that in the opinion of the investigator may interfere with the accurate evaluation of the subject's facial appearance.
9. Received any investigational drug or procedure within 28 days of the baseline visit or is scheduled to receive an investigational drug (other than the study products) or procedure during the study.
10. Currently using any medication that in the opinion of the investigator may affect the evaluation of the study products or place the subject at undue risk (including but not limited to asthma medications, oral steroids, rifampin, anticonvulsants, and St John's wart).
11. Has a history of known or suspected intolerance to any of the ingredients of the study products (ie, benzoyl peroxide).
12. Considered unable or unlikely to attend the necessary visits.
13. Live in the same household as currently enrolled subjects.
14. Employee of the investigator, a contract research organization, or Stiefel Laboratories who is involved in the study, or an immediate family member (partner, offspring, parents, siblings or sibling's offspring) of an employee involved in the study.

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09-01; Primary Completion 2010-01-01 (Actual); Study Completion 2010-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114550 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 participants were enrolled to an evaluator-blinded, split-face study of acne, which was conducted at two centers in United States from 08 September 2009 to 25 January 2010.
Pre-assignment Details: Same 20 participants were used in the split face study for the 2 interventions namely MaxClarity and Proactiv carried out in a single period.
Groups:
- MAXCLARITY II + PROACTIV: This was a split face study, wherein the participants, each morning washed their face with MaxClarity II foam cleanser on 1 side of the face and Proactive renewing cleanser on the other side of the face. The face was patted dry the MaxClarity II foam treatment was applied to the MaxClarity II side of the face and on the proactive side, the participant applied the Revitalizing toner and then the Repairing lotion. The same was repeated in the evening, where the participants washed their face with MaxClarity II foam cleanser on 1 side and Proactiv renewing cleanser on the other side of the face. On the Proactiv side, the participant will apply the Revitalizing toner and then the Repairing lotion.
Period: Overall Study
Arm/Group | MAXCLARITY II + PROACTIV
Started | 20
Completed | 18
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | MAXCLARITY II + PROACTIV
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.5 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black | 6
  White | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Inflammatory Lesion (IL), Non-inflammatory Lesion (NIL), and Total Lesion (TL) Counts From Baseline (BL) (Day 1) to Week (Wk) 8.
Description: This was an efficacy variable. An expert grader evaluated each side of the face (included forehead, cheeks and chin), the left and the right side, for IL (presence of papules and pustules), NIL (presence of open and closed comedones) and the TLs. The mouth, nose, periocular area, nasogenian, and superior and inferior eyelids were excluded. The evaluator was also blinded. BL was defined as Day 1. The percent change was calculated as the value at Wk 8 minus the value at BL.
Time Frame: BL (Day 1) and Wk 8
Population: The Intent to treat (ITT) analysis set included data from all randomized participants who received the study drug. The number of participants available at that particular time point were used for analysis.
Measure: Mean (Standard Deviation); unit: percent change in lesion count
Groups:
- MAXCLARITY II: MAXCLARITY II (2.5% benzyl peroxide [BPO]) foam cleanser and foam treatment, 0.5% salicylic acid toner foam were used in this arm, both morning and evening for 8-Wks. The participants in the morning washed their face with MaxClarity II foam cleanser, on 1 side of the face (the side of face, where no proactive cleanser and revitalizing toner were used) . The face was patted dry, post which MaxClarity II foam treatment was applied to the MaxClarity II side of the face. The same was repeated in the evening. This was a split face study.
- PROACTIV: Proactive renewing cleanser and revitalizing toner and the repairing lotion were used both morning and evening for 8-Wk, for the same participant, from Maxclarity II arm, on the other side. The same participants from the Maxclarity II arm, in the morning washed their face with Proactive renewing cleanser on the other side of the face. The face was patted dry, post which revitalizing toner and then the repairing lotion on the same side cleansed with the proactive cleanser. The same was repeated in the evening. This was a split face study.
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 18 | 18
percent change in lesion count
  Percent change, IL count | -55.93 (32.72) | -52.64 (29.23)
  Percent change, NIL count | -37.97 (38.72) | -45.66 (23.05)
  Percent change in TL count | -45.46 (27.24) | -47.69 (21.92)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Percent change for IL count for MAXCLARITY II Vs PROACTIV at Wk 8; Test type: Superiority or Other; p = 0.6779, t-test, 2 sided; Mean Difference (Net) = -3.29, Standard Deviation 32.98
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; Percent change for NIL count for MAXCLARITY II Vs PROACTIV at Wk 8; Test type: Superiority or Other; p = 0.2847, t-test, 2 sided; Median Difference (Net) = 7.68, Standard Deviation 29.51
Statistical Analysis 3: Comparison: MAXCLARITY II vs PROACTIV; Percent change for TL count for MAXCLARITY II Vs PROACTIV at Wk 8; Test type: Superiority or Other; p = 0.6894, t-test, 2 sided; Median Difference (Net) = 2.24, Standard Deviation 23.35

2. Secondary Outcome: Mean Percent Change in IL Count From BL (Day 1) to Wks 1, 2 and 4
Description: This was an efficacy variable. An expert grader (blinded) evaluated the left and the right side of the face extending from the hairline to the mandible (included forehead, cheeks and chin). The evaluator assessed the IL by counting the number of papules and pustules. The mouth, nose, periocular area, nasogenian, and superior and inferior eyelids were excluded. BL was defined as Day 1. The percent change was calculated as the percent value (count of IL) at each individual visit (percent value at wk 1, 2 and 4) minus the value at BL respectively.
Time Frame: BL (Day1) to Wks 1, 2 and 4
Population: ITT used. Only those participants available at the specified time points were analyzed (re presented by n=x, x in the category titles).
Measure: Mean (Standard Deviation); unit: percent change in lesion count
Groups:
- MAXCLARITY II: MAXCLARITY II (2.5% BPO) foam cleanser and foam treatment, 0.5% salicylic acid toner foam were used in this arm, both morning and evening for 8-Wk. The participants in the morning washed their face with MaxClarity II foam cleanser, on 1 side of the face (side of face, where no proactive cleanser and revitalizing toner were used) . The face was patted dry, post which MaxClarity II foam treatment was applied to the MaxClarity II side of the face. The same was repeated in the evening. This was a split face study.
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
percent change in lesion count
  Percent change, IL count, BL to Wk 1: number analyzed (Participants) | 20 | 19
  Percent change, IL count, BL to Wk 1 | -17.56 (33.63) | -19.93 (26.39)
  Percent change, IL count, BL to Wk 2: number analyzed (Participants) | 19 | 19
  Percent change, IL count, BL to Wk 2 | -35.64 (37.66) | -31.64 (30.06)
  Percent change, IL count, BL to Wk 4: number analyzed (Participants) | 19 | 19
  Percent change, IL count, BL to Wk 4 | -21.35 (63.62) | -44.99 (37.85)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Percent change for MAXCLARITY II Vs PROACTIV: IL count, BL to Wk 1 (within group); Test type: Superiority or Other; p = 0.9909, Signed Rank; Mean Difference (Net) = 2.38, Standard Deviation 50.10
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; IL count for MAXCLARITY II Vs PROACTIV- BL to Wk 2 (within group); Test type: Superiority or Other; p = 0.6671, t-test, 2 sided; Median Difference (Net) = -4.0, Standard Deviation 39.91
Statistical Analysis 3: Comparison: MAXCLARITY II vs PROACTIV; Percent change for MAXCLARITY II Vs PROACTIV: IL count, BL to Wk 4 (within group); Test type: Superiority or Other; p = 0.0632, t-test, 2 sided; Median Difference (Net) = 23.64, Standard Deviation 52.05

3. Secondary Outcome: Mean Percent Change in NIL Count From BL (Day 1) to Wks 1, 2 and 4
Description: This was an efficacy variable. An expert grader (blinded) evaluated the left and the right side of the face extending from the hairline to the mandible (included forehead, cheeks and chin). The evaluator assessed the NIL by the presence of open and closed comedones. The mouth, nose, periocular area, nasogenian, and superior and inferior eyelids were excluded. BL was defined as Day 1. The percent change was calculated as the percent value (count of NIL) at each individual visit (percent value at Wk 1, 2 and 4) minus the value at BL respectively.
Time Frame: BL (Day 1) to Wks 1, 2 and 4
Population: ITT population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: percent change in lesion count
Groups:
- MAXCLARITY II: MAXCLARITY II (2.5% BPO) foam cleanser and foam treatment, 0.5% salicylic acid toner foam were used in this arm, both morning and evening for 8-Wks. The participants in the morning washed their face with MaxClarity II foam cleanser, on 1 side of the face (side of face, where no proactive cleanser and revitalizing toner were used) . The face was patted dry, post which MaxClarity II foam treatment was applied to the MaxClarity II side of the face. The same was repeated in the evening. This was a split face study.
- PROACTIV: Proactive renewing cleanser and revitalizing toner and the repairing lotion were used both morning and evening for 8-Wks, for the same participant, from Maxclarity II arm, on the other side. The same participants from the Maxclarity II arm, in the morning washed their face with Proactive renewing cleanser on the other side of the face. The face was patted dry, post which revitalizing toner and then the repairing lotion on the same side cleansed with the proactive cleanser. The same was repeated in the evening. This was a split face study.
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
percent change in lesion count
  Percent change, NIL count, BL to Wk 1 | -3.92 (32.71) | -7.13 (25.91)
  Percent change, NIL count, BL to Wk 2: number analyzed (Participants) | 19 | 19
  Percent change, NIL count, BL to Wk 2 | -24.12 (37.73) | -21.07 (26.17)
  Percent change, NIL count, BL to Wk 4: number analyzed (Participants) | 19 | 19
  Percent change, NIL count, BL to Wk 4 | -30.26 (38.48) | -37.76 (22.65)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Percent change for MAXCLARITY II Vs PROACTIV: NIL count, BL to Wk 1 (within group); Test type: Superiority or Other; p = 0.7385, t-test, 2 sided; Mean Difference (Net) = 3.20, Standard Deviation 42.31
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; Percent change for MAXCLARITY II Vs PROACTIV: NIL count, BL to Wk 2 (within group); Test type: Superiority or Other; p = 0.7296, t-test, 2 sided; Mean Difference (Net) = -3.04, Standard Deviation 37.77
Statistical Analysis 3: Comparison: MAXCLARITY II vs PROACTIV; Percent change for MAXCLARITY II Vs PROACTIV: NIL count, BL to Wk 4 (within group); Test type: Superiority or Other; p = 0.3774, t-test, 2 sided; Mean Difference (Final Values) = 7.50, Standard Deviation 36.11

4. Secondary Outcome: Mean Percent Change in TL Count From BL (Day 1) to Wks 1, 2 and 4
Description: This was an efficacy variable. An expert grader (blinded) evaluated the left and the right side of the face extending from the hairline to the mandible (included forehead, cheeks and chin). The evaluator assessed the total lesions by the sum of both inflammatory and non-inflammatory lesions on each side (left side and right side). The mouth, nose, periocular area, nasogenian, and superior and inferior eyelids were excluded. BL was defined as Day 1. The percent change was calculated as the percent value (count of total lesions) at each individual visit (percent value at Wks 1, 2 and 4) minus the value at baseline respectively.
Time Frame: BL (Day 1) to Wks 1, 2 and 4
Population: ITT population. Only those participants available at the specified time points we re analyze d (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: percent change in lesion count
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
percent change in lesion count
  Percent change, in TL count, BL to Wk 1 | -11.34 (21.84) | -13.36 (19.07)
  Percent change, in TL count, BL to Wk 2: number analyzed (Participants) | 19 | 19
  Percent change, in TL count, BL to Wk 2 | -31.94 (27.86) | -26.19 (20.23)
  Percent change, in TL count, BL to Wk 4: number analyzed (Participants) | 19 | 19
  Percent change, in TL count, BL to Wk 4 | -34.17 (28.06) | -41.17 (20.23)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Percent change for MAXCLARITY II Vs PROACTIV: TL count, BL to Wk 1 (within group); Test type: Superiority or Other; p = 0.7634, t-test, 2 sided; Mean Difference (Net) = 2.02, Standard Deviation 29.53
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; Percent change for MAXCLARITY II Vs PROACTIV: TL count, BL to Wk 2 (within group); Test type: Superiority or Other; p = 0.4087, t-test, 2 sided; Mean Difference (Net) = -5.75, Standard Deviation 29.61
Statistical Analysis 3: Comparison: MAXCLARITY II vs PROACTIV; Percent change for MAXCLARITY II Vs PROACTIV: TL count, BL to Wk 4 (within group); Test type: Superiority or Other; p = 0.2455, t-test, 2 sided; Mean Difference (Net) = 7.00, Standard Deviation 25.40

5. Secondary Outcome: Mean Change in Investigator's Static Global Assessment (ISGA) From BL (Day 1) to Wks 1, 2, 4 and 8.
Description: The evaluator (blinded) evaluated the acne severity of the participants' face using the ISGA scale ranging from 0 to 5. The grading was 0= Clear, skin with no IL or NILs; 1= Almost clear, rare NILs with no more than one small IL ; 2= Mild, some NILs with no more than few ILs (papules/pustules only, no nodular lesions); 3= Moderate Upto many NILs and may have some ILs but no more than one small nodular lesion ; 4= Severe, Upto many NILs and ILs but no more than a few nodular lesions; 5= Very severe, many NILS and ILs more than a few nodular lesions, may have cystic lesions. Thus higher score indicated severity of the disease. BL was defined as Day 1. The mean change was calculated as value at each visit (Wks 1,2,4 and 8) minus the value at BL respectively.
Time Frame: BL (Day 1) to Wks 1, 2, 4 and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
units on scale
  Change, in ISGA from BL to Wk 1 | -0.10 (0.31) | -0.05 (0.39)
  Change, in ISGA from BL to Wk 2: number analyzed (Participants) | 19 | 19
  Change, in ISGA from BL to Wk 2 | -0.47 (0.61) | -0.21 (0.54)
  Change, in ISGA from BL to Wk 4: number analyzed (Participants) | 19 | 19
  Change, in ISGA from BL to Wk 4 | -0.53 (0.51) | -0.42 (0.61)
  Change, in ISGA from BL to Wk 8: number analyzed (Participants) | 18 | 18
  Change, in ISGA from BL to Wk 8 | -0.39 (0.61) | -0.39 (0.61)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Change, in ISGA for MAXCLARITY II Vs PROACTIV: from BL to Wk 1 (within group); Test type: Superiority or Other; p = 1.0000, Signed Rank; Mean Difference (Net) = -0.05, Standard Deviation 0.39
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; Change, in ISGA for MAXCLARITY II Vs PROACTIV: from BL to Wk 2 (within group); Test type: Superiority or Other; p = 0.1250, Signed Rank; Mean Difference (Net) = -0.26, Standard Deviation 0.56
Statistical Analysis 3: Comparison: MAXCLARITY II vs PROACTIV; Change, in ISGA for MAXCLARITY II Vs PROACTIV: from BL to Wk 4 (within group); Test type: Superiority or Other; p = 0.6250, Signed Rank; Mean Difference (Net) = -0.11, Standard Deviation 0.46
Statistical Analysis 4: Comparison: MAXCLARITY II vs PROACTIV; Change, in ISGA for MAXCLARITY II Vs PROACTIV: from BL to Wk 8 (within group); Test type: Superiority or Other; p = 1.0000, Signed Rank; Mean Difference (Net) = 0.00, Standard Deviation 0.59

6. Secondary Outcome: Mean Change in Each of the Evaluator Tolerability Assessments-Erythema
Description: This was a tolerability variable. The expert grader (blinded evaluator) assessed each left and right side of the face individually at each study visit. The areas on the face excluding nose, nasogenian, and superior and inferior eyelids were evaluated. The evaluator conducting the assessment for the participant remained blinded for the treatment assigned. Erythema is condition characterized by redness or rash on the skin. The assessment of the erythema was graded on 0 to 5 scale based on severity by the evaluator. 0=None, 1=Very minimal, 2=mild, 3= moderate, 4=severe, and 5= Very severe. Thus higher score indicated severity of the disease. BL was defined as Day 1. The mean change was calculated as value at each individual visit (wk 1,2,4 and 8) minus the value at BL respectively. The change from BL was '0' for Wk 4 and Wk 8, and hence statistical analysis was not done.
Time Frame: BL (Day 1) to Wks 1, 2, 4 and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Groups:
- MAXCLARITY II: MAXCLARITY II (2.5% BPO) foam cleanser and foam treatment, 0.5% salicylic acid toner foam were used in this arm, both morning and evening for 8-weeks (Wk). The participants in the morning washed their face with MaxClarity II foam cleanser, on 1 side of the face (side of face, where no proactive cleanser and revitalizing toner were used) . The face was patted dry, post which MaxClarity II foam treatment was applied to the MaxClarity II side of the face. The same was repeated in the evening. This was a split face study.
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
units on scale
  Erythema; Change from BL to Wk 1 | 0.05 (0.51) | -0.05 (0.22)
  Erythema; Change from BL to Wk 2: number analyzed (Participants) | 19 | 19
  Erythema; Change from BL to Wk 2 | -0.05 (0.23) | -0.11 (0.32)
  Erythema; Change from BL to Wk 4: number analyzed (Participants) | 19 | 19
  Erythema; Change from BL to Wk 4 | 0.05 (0.40) | 0.05 (0.40)
  Erythema; Change from BL to Wk 8: number analyzed (Participants) | 18 | 18
  Erythema; Change from BL to Wk 8 | 0.06 (0.42) | 0.06 (0.42)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Change, in Erythema for MAXCLARITY II Vs PROACTIV: from BL to Wk 1 (within group); Test type: Superiority or Other; p = 1.0000, Signed Rank; Mean Difference (Net) = 0.10, Standard Deviation 0.45
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; Change, in Erythema for MAXCLARITY II Vs PROACTIV: from BL to Wk 2 (within group); Test type: Superiority or Other; p = 1.0000, Signed Rank; Signed Rank = 0.05, Standard Deviation 0.23

7. Secondary Outcome: Mean Change in Each of the Evaluator Tolerability Assessments-Dryness
Description: This was a tolerability variable. The expert grader (blinded evaluator) assessed each left and right side of the face individually at each study visit. The areas on the face excluding nose, nasogenian, and superior and inferior eyelids were evaluated. The evaluator conducting the assessment for the participant remained blinded for the treatment assigned. The assessment of the dryness was graded on 0 to 5 scale based on severity by the evaluator. 0=None, 1=Very minimal, 2=mild, 3= moderate, 4=severe, and 5= Very severe. Thus higher score indicated more severity. BL was defined as Day 1. The mean change was calculated as value at each individual visit (Wk 1,2,4 and 8) minus the value at baseline respectively. The change from BL was '0' for Wk 2, Wk 4, and Wk 8 and hence statistical analysis was not done.
Time Frame: BL (Day 1) to Wks 1, 2, 4 and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
units on scale
  Dryness; Change from BL to Wk 1 | 0.15 (0.49) | 0.10 (0.45)
  Dryness; Change from BL to Wk 2: number analyzed (Participants) | 19 | 19
  Dryness; Change from BL to Wk 2 | 0.00 (0.00) | 0.00 (0.00)
  Dryness; Change from BL to Wk 4: number analyzed (Participants) | 19 | 19
  Dryness; Change from BL to Wk 4 | 0.05 (0.23) | 0.00 (0.00)
  Dryness; Change from BL to Wk 8: number analyzed (Participants) | 18 | 18
  Dryness; Change from BL to Wk 8 | 0.11 (0.32) | 0.11 (0.32)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Change, in Dryness for MAXCLARITY II Vs PROACTIV: from BL to Wk 1 (within group); Test type: Superiority or Other; p = 1.00, Signed Rank; Mean Difference (Net) = 0.05, Standard Deviation 0.22
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; Change, in Dryness for MAXCLARITY II Vs PROACTIV: from BL to Wk 4 (within group); Test type: Superiority or Other; p = 1.0000, Signed rank; Mean Difference (Net) = 0.05, Standard Deviation 0.23

8. Secondary Outcome: Mean Change in Each of the Evaluator Tolerability Assessments-Peeling
Description: This was a tolerability variable. The expert grader (blinded evaluator) assessed each left and right side of the face individually at each study visit. The areas on the face excluding nose, nasogenian, and superior and inferior eyelids were evaluated. The evaluator conducting the assessment for the participant remained blinded for the treatment assigned. The assessment of the peeling was graded on 0 to 5 scale based on severity by the evaluator. 0=None, 1=Very minimal, 2=mild, 3= moderate, 4=severe, and 5= Very severe. Thus higher score indicated more severity. BL was defined as Day 1. The mean change was calculated as value at each individual visit (Wk 1,2,4 and 8) minus the value at BL respectively. The change from BL was '0' for Wk (1, 4 and 8) and hence statistical analysis was not done.
Time Frame: BL (Day 1) to Wks 1, 2, 4 and 8
Population: ITT population. Only those participants available at the specified time points were analyze d (represented by n=x, x in the category titles).
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
units on scale
  Peeling; Change from BL to Wk 1 | 0.00 (0.00) | 0.00 (0.00)
  Peeling; Change from BL to Wk 2: number analyzed (Participants) | 19 | 19
  Peeling; Change from BL to Wk 2 | 0.00 (0.00) | 0.11 (0.46)
  Peeling; Change from BL to Wk 4: number analyzed (Participants) | 19 | 19
  Peeling; Change from BL to Wk 4 | 0.00 (0.00) | 0.00 (0.00)
  Peeling; Change from BL to Wk 8: number analyzed (Participants) | 18 | 18
  Peeling; Change from BL to Wk 8 | 0.00 (0.00) | 0.00 (0.00)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Change, in Peeling, for MAXCLARITY II Vs PROACTIV: from BL to Wk 2 (within group); Test type: Superiority or Other; p = 1.0000, Signed rank; Mean Difference (Net) = -0.11, Standard Deviation 0.46

9. Secondary Outcome: Mean Change in Each of the Participant Tolerability Assessments-Redness
Description: This was a tolerability variable, where the participants were instructed to individually assess the right and the left side of the face to indicate the severity that they had experienced during the time period from their last visit for redness. The area on the face was assessed excluding the excluding nose, nasogenian, and superior and inferior eyelids. The assessment of the redness was graded on 0 to 5 scale based on severity by the participant. 0=None, 1=Very minimal, 2=mild, 3= moderate, 4=severe, and 5= Very severe. Thus higher score indicated more severity. BL was defined as Day 1. The mean change was calculated as value at each individual visit (Wks 1,2,4 and 8) minus the value at BL respectively.
Time Frame: BL (Day 1) to Wks 1, 2, 4 and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
units on scale
  Redness; Change from BL to Wk 1 | 0.50 (1.00) | 0.35 (0.81)
  Redness; Change from BL to Wk 2: number analyzed (Participants) | 19 | 19
  Redness; Change from BL to Wk 2 | 0.37 (1.01) | 0.21 (0.79)
  Redness; Change from BL to Wk 4: number analyzed (Participants) | 18 | 18
  Redness; Change from BL to Wk 4 | 0.72 (1.13) | 0.56 (0.86)
  Redness; Change from BL to Wk 8: number analyzed (Participants) | 18 | 18
  Redness; Change from BL to Wk 8 | 0.61 (1.14) | 0.28 (0.75)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Change, in Redness for MAXCLARITY II Vs PROACTIV: from BL to Wk 1 (within group); Test type: Superiority or Other; p = 0.5313, Signed Rank; Mean Difference (Net) = 0.15, Standard Deviation 0.67
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; Change, in Redness for MAXCLARITY II Vs PROACTIV: from BL to Wk 2 (within group); Test type: Superiority or Other; p = 0.5000, Signed Rank; Median Difference (Net) = 0.16, Standard Deviation 0.60
Statistical Analysis 3: Comparison: MAXCLARITY II vs PROACTIV; Change, in Redness for MAXCLARITY II Vs PROACTIV: from BL to Wk 4 (within group); Test type: Superiority or Other; p = 0.7500, Signed Rank; Mean Difference (Net) = 0.17, Standard Deviation 0.86
Statistical Analysis 4: Comparison: MAXCLARITY II vs PROACTIV; Change, in Redness for MAXCLARITY II Vs PROACTIV: from BL to Wk 8 (within group); Test type: Superiority or Other; p = 0.2500, Signed rank; Mean Difference (Net) = 0.33, Standard Deviation 0.84

10. Secondary Outcome: Mean Change in Each of the Participant Assessments of Tolerability-Dryness
Description: This was a tolerability variable, where the participants were instructed to individually assess the right and the left side of the face to indicate the severity that they had experienced during the time period from their last visit for dryness. The area on the face was assessed excluding the excluding nose, nasogenian, and superior and inferior eyelids. The assessment of the dryness was graded on 0 to 5 scale based on severity by the participant. 0=None, 1=Very minimal, 2=mild, 3= moderate, 4=severe, and 5= Very severe. Thus higher score indicated severity of the disease. BL was defined as Day 1. The mean change was calculated as value at each individual visit (Wks 1,2,4 and 8) minus the value at BL respectively.
Time Frame: BL (Day 1) to Wks 1, 2, 4 and 8
Population: ITT population . Only those participants available at the specified time points we re analyze d (represented by n=x, x in the category titles).
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
units on scale
  Dryness; Change from BL to Wk 1 | 1.20 (1.24) | 0.90 (1.07)
  Dryness; Change from BL to Wk 2: number analyzed (Participants) | 19 | 19
  Dryness; Change from BL to Wk 2 | 1.05 (1.39) | 0.68 (1.16)
  Dryness; Change from BL to Wk 4: number analyzed (Participants) | 18 | 18
  Dryness; Change from BL to Wk 4 | 1.33 (1.14) | 1.06 (1.00)
  Dryness; Change from BL to Wk 8: number analyzed (Participants) | 18 | 18
  Dryness; Change from BL to Wk 8 | 1.33 (1.24) | 1.11 (1.02)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Change, in Dryness for MAXCLARITY II Vs PROACTIV: from BL to Wk 1 (within group); Test type: Superiority or Other; p = 0.2131, Signed Rank); Mean Difference (Net) = 0.30, Standard Deviation 0.86
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; Change, in Dryness for MAXCLARITY II Vs PROACTIV: from BL to Wk 2 (within group); Test type: Superiority or Other; p = 0.2656, Signed Rank; Mean Difference (Net) = 0.37, Standard Deviation 1.16
Statistical Analysis 3: Comparison: MAXCLARITY II vs PROACTIV; Change, in Dryness for MAXCLARITY II Vs PROACTIV: from BL to Wk 4 (within group); Test type: Superiority or Other; p = 0.2344, Signed Rank; Mean Difference (Net) = 0.28, Standard Deviation 0.75
Statistical Analysis 4: Comparison: MAXCLARITY II vs PROACTIV; Change, in Dryness for MAXCLARITY II Vs PROACTIV: from BL to Wk 8 (within group); Test type: Superiority or Other; p = 0.3594, Signed Rank; Mean Difference (Net) = 0.22, Standard Deviation 0.73

11. Secondary Outcome: Mean Change in Each of the Participant Assessments of Tolerability-Burning
Description: This was a tolerability variable, where the participants were instructed to individually assess the right and the left side of the face to indicate the severity that they had experienced during the time period from their last visit for burning. The area on the face was assessed excluding nose, nasogenian, and superior and inferior eyelids. The assessment of the burning was graded on 0 to 5 scale based on severity by the participant; 0=None, 1=Very minimal, 2=mild, 3= moderate, 4=severe, and 5= Very severe. Thus higher score indicated more severity. BL was defined as Day 1. The mean change was calculated as value at each individual visit (Wks 1, 2, 4 and 8) minus the value at BL respectively.
Time Frame: BL (Day 1) to Wks 1,2, 4 and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
units on scale
  Burning; Change from BL to Wk 1 | 0.95 (1.28) | 0.75 (0.85)
  Burning; Change from BL to Wk 2: number analyzed (Participants) | 19 | 19
  Burning; Change from BL to Wk 2 | 0.84 (1.17) | 0.58 (0.84)
  Burning; Change from BL to Wk 4: number analyzed (Participants) | 18 | 18
  Burning; Change from BL to Wk 4 | 1.00 (1.08) | 0.44 (0.62)
  Burning; Change from BL to Wk 8: number analyzed (Participants) | 18 | 20
  Burning; Change from BL to Wk 8 | 0.83 (1.34) | 0.44 (0.70)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Change, in Burning for MAXCLARITY II Vs PROACTIV: from BL to Wk 1 (within group); Test type: Superiority or Other; p = 0.6172, Signed Rank; Mean Difference (Net) = 0.20, Standard Deviation 1.32
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; Change, in Burning for MAXCLARITY II Vs PROACTIV: from BL to Wk 2 (within group); Test type: Superiority or Other; p = 0.3984, Signed Rank; Mean Difference (Net) = 0.26, Standard Deviation 0.93
Statistical Analysis 3: Comparison: MAXCLARITY II vs PROACTIV; Change, in Burning for MAXCLARITY II Vs PROACTIV: from BL to Wk 4 (within group); Test type: Superiority or Other; p = 0.0781, Signed Rank; Mean Difference (Net) = 0.56, Standard Deviation 1.10
Statistical Analysis 4: Comparison: MAXCLARITY II vs PROACTIV; Change, in Burning for MAXCLARITY II Vs PROACTIV: from BL to Wk 8 (within group); Test type: Superiority or Other; p = 0.3750, Signed Rank; Mean Difference (Net) = 0.39, Standard Deviation 1.24

12. Secondary Outcome: Mean Change in Each of the Participant Assessments of Tolerability-Itching
Description: This was a tolerability variable, where the participants were instructed to individually assess the right and the left side of the face to indicate the severity that they had experienced during the time period from their last visit for itching. The area on the face was assessed excluding nose, nasogenian, and superior and inferior eyelids. The assessment of the itching was graded on 0 to 5 scale based on severity by the participant; 0=None, 1=Very minimal, 2=mild, 3= moderate, 4=severe, and 5= Very severe. Thus higher score indicated more severity. BL was defined as Day 1. The mean change was calculated as value at each individual visit (Wks 1,2,4 and 8) minus the value at BL respectively.
Time Frame: BL (Day 1) to Wks 1, 2, 4 and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
units on scale
  Itching; Change from BL to Wk 1 | 0.20 (0.62) | 0.20 (0.77)
  Itching; Change from BL to Wk 2: number analyzed (Participants) | 19 | 19
  Itching; Change from BL to Wk 2 | 0.37 (1.01) | 0.05 (0.62)
  Itching; Change from BL to Wk 4: number analyzed (Participants) | 18 | 18
  Itching; Change from BL to Wk 4 | 0.33 (0.97) | 0.06 (0.24)
  Itching; Change from BL to Wk 8: number analyzed (Participants) | 18 | 18
  Itching; Change from BL to Wk 8 | 0.28 (0.57) | 0.11 (0.58)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Change, in Itching for MAXCLARITY II Vs PROACTIV: from BL to Wk 1 (within group); Test type: Superiority or Other; p = 1.0000, [Signed Rank]; Median Difference (Net) = 0.00, Standard Deviation 0.46
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; Change, in Itching for MAXCLARITY II Vs PROACTIV: from BL to Wk 2 (within group); Test type: Superiority or Other; p = 0.0625, Signed Rank; Mean Difference (Net) = 0.32, Standard Deviation 0.58
Statistical Analysis 3: Comparison: MAXCLARITY II vs PROACTIV; Change, in Itching for MAXCLARITY II Vs PROACTIV: from BL to Wk 4 (within group); Test type: Superiority or Other; p = 0.2500, Signed Rank; Mean Difference (Net) = 0.28, Standard Deviation 0.75
Statistical Analysis 4: Comparison: MAXCLARITY II vs PROACTIV; Change, in Itching for MAXCLARITY II Vs PROACTIV: from BL to Wk 8 (within group); Test type: Superiority or Other; p = 0.2500, Signed Rank; Mean Difference (Net) = 0.17, Standard Deviation 0.38

13. Secondary Outcome: Mean Change in Each of the Participant Assessments of Tolerability-Scaling
Description: This was a tolerability variable, where the participants were instructed to individually assess the right and the left side of the face to indicate the severity that they had experienced during the time period from their last visit for scaling. The area on the face was assessed excluding nose, nasogenian, and superior and inferior eyelids. The assessment of the scaling was graded on 0 to 5 scale based on severity by the participant; 0=None, 1=Very minimal, 2=mild, 3= moderate, 4=severe, and 5= Very severe. Thus higher score indicated more severity. BL was defined as Day 1. The mean change was calculated as value at each individual visit (Wks 1,2,4 and 8) minus the value at BL respectively.
Time Frame: BL (Day 1) to Wks 1, 2, 4 and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | MAXCLARITY II | PROACTIV
Number analyzed (Participants) | 20 | 20
units on scale
  Scaling; Change from BL to Wk 1 | 0.40 (0.68) | 0.25 (0.55)
  Scaling; Change from BL to Wk 2: number analyzed (Participants) | 19 | 19
  Scaling; Change from BL to Wk 2 | 0.26 (0.81) | 0.16 (0.69)
  Scaling; Change from BL to Wk 4: number analyzed (Participants) | 18 | 18
  Scaling; Change from BL to Wk 4 | 0.56 (0.86) | 0.39 (0.78)
  Scaling; Change from BL to Wk 8: number analyzed (Participants) | 18 | 18
  Scaling; Change from BL to Wk 8 | 0.83 (1.20) | 0.67 (1.14)
Statistical Analysis 1: Comparison: MAXCLARITY II vs PROACTIV; Change, in Scaling for MAXCLARITY II Vs PROACTIV: from BL to Wk 1 (within group); Test type: Superiority or Other; p = 0.5000, Signed Rank; Signed Rank = 0.15, Standard Deviation 0.59
Statistical Analysis 2: Comparison: MAXCLARITY II vs PROACTIV; Change, in Scaling for MAXCLARITY II Vs PROACTIV: from BL to Wk 2 (within group); Test type: Superiority or Other; p = 0.7500, Signed Rank; Signed Rank = 0.11, Standard Deviation 0.57
Statistical Analysis 3: Comparison: MAXCLARITY II vs PROACTIV; Change, in Scaling for MAXCLARITY II Vs PROACTIV: from BL to Wk 4 (within group); Test type: Superiority or Other; p = 0.4531, Signed Rank; Mean Difference (Net) = 0.17, Standard Deviation 0.62
Statistical Analysis 4: Comparison: MAXCLARITY II vs PROACTIV; Change, in Scaling for MAXCLARITY II Vs PROACTIV: from BL to Wk 8 (within group); Test type: Superiority or Other; p = 0.6250, Signed Rank; Mean Difference (Net) = 0.17, Standard Deviation 0.86

ADVERSE EVENTS:
Time Frame: From the informed consent taken to up to 4 months
Description: ITT Population. There were no treatment -related adverse events reported during the study, so the data has been reported as an overall, single arm; as the participants used were the same in each arm
Arm/Group | MAXCLARITY II + PROACTIV
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAXCLARITY II + PROACTIV (N=20)
Nasopharyngitis (Infections and infestations) | 3
Skin infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.